CLINICAL TRIAL: NCT03118323
Title: Patients' Willingness-to-pay of Endodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Göttingen (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Dr. med. dent., Dr. rer. medic., Dr. med. dent., University Medical Center Goettingen
Other Study IDs: WTP-Endodontic
Record Dates: First submitted 2017-04-12; First posted 2017-04-18 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Patient Preference
Keywords: willingness topay; WTP; health economic; preference-based measures
MeSH Terms: conditions — Patient Preference | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients in need of endodontic treatment: n = 200
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients are given a questionnaire with items related to personality and their willingness-to-pay for different treatment options.

SUMMARY:
The aim of the present study is to determine the monetary value of endodontic treatment (primary root canal treatment) compared to the alternative treatment options, such as extraction with or without subsequent insertion of a dental implant or placement of a fixed dental prosthesis.

DETAILED DESCRIPTION:
Endodontic treatment of teeth with irreversibly damaged pulp aim at the long-term preservation of the affected tooth. If contraindications are present and / or a patient refuse endodontic treatment, the extraction of the affected tooth is often necessary. The resulting tooth gap might be closed by inserting a dental implant or by placing a fixed dental prosthesis.

Prior studies have shown that patients' decisions in alternative treatment options depend on a variety of factors. Studies on the willingness-to-pay (WTP) are used to compare the monetary value of different therapy procedures.

ELIGIBILITY:
Participants are selected by consecutive patient sampling (total n = 200).

Inclusion Criteria:

* Patients who are in need of an primary root canal treatment and who are able to give written consent

Exclusion Criteria:

* Non-fulfillment of the inclusion criteria
* Lack of capacity to consent
* No German language skills in written and spoken language
* Age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Department of Preventive Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
  * Department of Operative and Preventive Dentistry, Charité - Universitätsmedizin Berlin, Germany
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-08 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Completion of a questionnaire | 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Principal Investigator — Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Germany
Locations (2):
- Germany (2):
  - University Medical Center Göttingen, Dept. of Preventive Dentistry, Periodontology and Cariology, Göttingen, Lower Saxony
  - Charité - Universitätsmedizin Berlin, Dept. of Operative and Preventive Dentistry, Berlin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ernst J, Brahler E, Weissflog G. [Patient involvement in medical decision making--an overview on patient preferences and impacting factors]. Gesundheitswesen. 2014 Apr;76(4):187-92. doi: 10.1055/s-0033-1361150. Epub 2014 Jan 9. German. PMID 24408309
- [Background] Gelberg L, Andersen RM, Leake BD. The Behavioral Model for Vulnerable Populations: application to medical care use and outcomes for homeless people. Health Serv Res. 2000 Feb;34(6):1273-302. PMID 10654830
- [Background] Herrera A, Martin J, Perez F, Bonafe E, Reis A, Dourado AL, Fernandez E. Is personality relevant in the choice of bleaching? Clin Oral Investig. 2016 Nov;20(8):2105-2111. doi: 10.1007/s00784-015-1701-3. Epub 2016 Jan 11. PMID 26750134
- [Background] Vernazza CR, Steele JG, Whitworth JM, Wildman JR, Donaldson C. Factors affecting direction and strength of patient preferences for treatment of molar teeth with nonvital pulps. Int Endod J. 2015 Dec;48(12):1137-46. doi: 10.1111/iej.12413. Epub 2014 Dec 10. PMID 25400281